CLINICAL TRIAL: NCT01914484
Title: A PHASE I/II, MULTI-CENTRE, TRIAL OF RUXOLITINIB THERAPY IN COMBINATION WITH NILOTINIB IN PATIENTS WITH PHILADELPHIA POSITIVE CHRONIC MYELOID LEUKEMIA OR ACUTE LYMPHOBLASTIC LEUKEMIA WHO HAVE FAILED TYROSINE KINASE INHIBITOR THERAPY
Brief Title: Phase I/II Study of Nilotinib/Ruxolitinb Therapy for TKI Resistant Ph-Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107ACA06T; OZM-051 (Other: Ozmosis)
Record Dates: First submitted 2013-07-28; First posted 2013-08-02 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Chronic Phase Chronic Myeloid Leukemia; Accelerated Phase Chronic Myeloid Leukemia; Blastic Phase Chronic Myeloid Leukemia; Philadelphia Positive Acute Lymphoblastic Leukemia; Resistant to Tyrosine Kinase Inhibitor Therapy
Keywords: tyrosine kinase inhibitor resistance; chronic myeloid leukemia; acute lymphoblastic leukemia; nilotinib; ruxolitinib
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib with Ruxolitinib (Experimental): Nilotinib: Given that recommended dose of Nilotinib for imatinib failed CML patients is 400mg twice daily, Nilotinib dose will remain fixed at 400mg bid throughout the cycles.
  Ruxolitinib: In the phase I part of the study, dose escalation will follow a 3+3 study design. Dose modifications will not occur, as the purpose of this study is to determine the maximum tolerated dose. Ruxolitinib will be given at one of 3 fixed dose levels for the duration of their treatment, either 10mg twice daily, 15mg twice daily or 20mg twice daily.
  Interventions: Drug: Nilotinib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib dose will remain fixed at 400mg bid throughout the cycles. BCR-ABL kinase inhibitor
  Other Names: Tasigna
Drug: Ruxolitinib — In the phase I part of the study, dose escalation will follow a 3+3 study design at either of 3 fixed dose levels (10 mg bid, 15 mg bid or 20 mg bid).
  No intra-patient dose-escalation will occur. JAK inhibitor
  Other Names: INCB018424; Jakavi

SUMMARY:
This is the study to test combination regimen of Nilotinib and Ruxolitinib therapy for the treatment of patients with Philadelphia positive chronic myeloid leukemia (CML) or acute lymphoblastic leukemia (ALL) who is resistant to multiple tyrosine kinase inhibitor therapies with BCR-ABL kinase inhibition activity. Ruxolitinib is a tyrosine kinase inhibitor blocking alternative pathway independent of BCR-ABL mediated pathway, thus having a potential to overcome tyrosine kinase inhibitor resistance in Philadelphia positive CML or ALL patients. Phase I study will be conducted to define a recommended phase II dose (RPTD) and phase II study will examine the hypothesis that combinational approach will increase response rate of resistant CML/ALL patients, thus evaluating efficacy of the combination regimen.

DETAILED DESCRIPTION:
The purpose of this study is to find out if multiple tyrosine kinase inhibitor resistant chronic myeloid leukemia (CML) or acute lymphoblastic leukemia (ALL) can be treated with combination approach of Nilotinib with Ruxolitinib which may block alternative pathway besides BCR-ABL kinase inhibition in Ph positive leukemia, esp against JAK2-STAT5 pathway. First step is to define the dose of Ruxolitinib with fixed dose of Nilotinib which had been approved at the dose of 400mg bid for imatinib failed CML.

During phase I part of the study,dose escalations will be decided on the basis of DLTs observed hence the exact sample size could not be predicted with certainty but will range between 9-12 patients. Three patients will be enrolled per dose level. Accordingly 9 patients are expected to be enrolled. If a DLT is observed, 3 more patients will be enrolled at the dose level in which the DLT occurred.

The study will be conducted at multiple sites across Canada and enrollment will be competitive. Once 3 patients are enrolled in a cohort, that dose level will be closed to enrollment until safety assessment of the 3 subjects is performed at the end of cycle 1. This procedure will be performed for each dosing cohort. Patients will be assigned to a dose level based on authorization from the sponsor in collaboration with Ozmosis Research Inc.

For the phase II part of the study, once the RPTD has been established in the phase I portion of this trial, the phase II will begin. The phase II portion will be a two-stage, single arm, unblinded study investigating the potential efficacy of the combination of Ruxolitinib and Nilotinib.

A maximum of 20 patients will be accrued in the phase II portion. Those patients treated in the phase I portion of this trial at the RPTD will be included in the analysis of the Phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have Chronic Myeloid Leukemia in any phase (CP, AP, or BP of any phenotype) or Ph+ Acute Lymphoblasic Leukemia. The confirmation of Ph+ chromosome can be substituted by the presence of BCR/ABL transcript by PCR test at diagnosis.
2. Patients must be previously treated with and resistant, or intolerant, to 2 or more lines of treatment including imatinib, dasatinib, or other investigational agent. Patient who have CML-CP who were previously treated with and resistant to only dasatinib are also included. At least 2 weeks must have elapsed from the last date of treatment to the first dose of study treatment. Patients who have received Nilotinib for more than 4 consecutive weeks will be excluded.
3. Must be ≥18 years old.
4. Provide written informed consent.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Minimum life expectancy of 3 months or more.
7. Adequate organ liver and renal functions:

   * Total bilirubin ≤ 1.5 x ULN. Does not apply to patients with isolated hyperbilirubinemia (e.g., Gilbert's Disease) of grade < 3;
   * Alanine aminotransferase (ALT) ≤ 2.5x ULN or or ≤ 5.0 x ULN if considered due to leukemia.
   * Creatinine ≤ 2.5 mg/dL.
   * Alkaline phosphatase ≤ 2.5 x ULN unless considered due to leukemia;
   * Serum lipase and amylase ≤ 1.5 x ULN
8. Normal serum levels ≥ LLN (lower limit of normal) or corrected to within normal limits with supplements, prior to the first dose of study medication, of potassium, magnesium and calcium;
9. Female patients of childbearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test within 2 weeks prior to enrollment. Male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. Acceptable methods of contraception are condoms, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post menopausal. Post menopausal is defined as at least 12 consecutive months without menses.
10. Ability and willingness to comply with study procedures and schedule, in the Investigator's opinion.

Exclusion Criteria:

1. Received Tyrosine Kinase Inhibitor therapy within 7 days prior to receiving the first dose of Ruxolitinib+Nilotinib, with the exception of patients who have previously received Nilotinib who must have stopped Nilotinib 4 weeks prior to receiving the first dose of Ruxolitinib+Nilotinib.

   Patients who have not recovered (> grade 1 by NCI CTCAE, v. 4.03) from AEs (except alopecia) due to agents previously administered.
2. Patients who received other therapies as follows:

   * For CP and AP patients:

   Received any of the following within 2 weeks prior to receiving first dose of Ruxolitinib + Nilotinib:
   * Hydroxyurea (within 7 days of first dose)
   * anagrelide
   * interferon
   * cytarabine
   * immunotherapy
   * any other cytotoxic chemotherapy, radiotherapy, or investigational therapy

     * For BP patients:

   Received any of the following within 2 weeks prior to receiving first dose of Ruxolitinib + Nilotinib:
   * chemotherapy other than hydroxyurea
   * anagrelide
   * interferon
   * cytarabine
   * immunotherapy
   * any other cytotoxic chemotherapy, radiotherapy, or investigational therapy

     * For Ph+ ALL patients:

   Received any of the following within 2 weeks prior to the first dose of Ruxolitinib+Nilotinib:
   * corticosteroids
   * vincristine
   * Hydroxyurea (within 7 days of first dose)
   * anagrelide
   * interferon
   * cytarabine
   * immunotherapy
   * any other cytotoxic chemotherapy, radiotherapy, or investigational therapy
3. Underwent autologous or allogeneic stem cell transplant within 60 days prior to receiving the first dose of Ruxolitinib+Nilotinib; any evidence of on-going graft versus-host disease (GVHD), or GVHD requiring immunosuppressive therapy.
4. Patients with any of the following:

   Have prolonged QT (QTc >450 ms) or take medications that are known to be associated with Torsades de Pointes, or potentially prolonging QT.

   Long QT syndrome or familiar history of long QT syndrome Persistent significant bradicardia (<50bpm) Experienced a myocardial infarction within 12 months of registration
5. Require concurrent treatment with immunosuppressive agents, other than corticosteroids prescribed for a short course of therapy.
6. Have previously been treated with Ruxolitinib.
7. Patients with CML CP are excluded if they are in MCyR.
8. Patients with CML AP, CML BP, or Ph+ ALL are excluded if they are in MCyR.
9. Have active central nervous system (CNS) disease as evidenced by cytology or pathology. History itself of CNS involvement is not exclusionary if CNS has been cleared with a documented negative lumbar puncture. In the absence of clinical CNS disease, lumbar puncture is not required.
10. Have significant or active cardiovascular disease or significant bleeding disorder unrelated to CML or Ph+ ALL.
11. Have a history of pancreatitis or alcohol abuse.
12. Have uncontrolled hypertriglyceridemia (triglycerides >450 mg/dL).
13. Have malabsorption syndrome or other gastrointestinal illness that could affect the absorption of the study drug.
14. Patients with inadequate bone marrow reserve within 2 weeks prior to start study drug as demonstrated by:

    * Absolute neutrophil count (ANC) that is ≤ 1000/µL.
    * Platelet count that is < 125,000/µL without the assistance of growth factors, thrombopoietic factors or platelet transfusions.
15. Patients with any history of platelet counts < 50,000/µL or ANC < 500/µL except during treatment for a myeloproliferative disorder or treatment with cytotoxic therapy for any other reason.
16. Patients with coagulation parameters (PT, PTT, INR) ≥ 1.5 ULN within 2 weeks prior to starting study drug.
17. Developed the T315I, T315A Y253H, E255K/V or F359C/V mutation after any TKI therapy.
18. Patients with HLA matched donor and eligible for allogeneic transplantation for CML treatment.
19. Patient being treated concurrently with any of the following prohibited medications:

    * JAK inhibitor
    * Any investigational medication other than the study drugs. Use of such medications within 14 days or 6 half-lives, whichever is longer, prior to the first dose of study drug is prohibited
    * Potent inducers and inhibitors of CYP3A4• Use of HU, interferon, thalidomide, busulfan, lenalidomide, anagrelide, is not permitted at any time beginning 28 days prior to the first Baseline assessment.
    * Hematopoietic growth factor receptor agonists (eg, erythropoietin (Epo), granulocyte colony stimulating factor (GCSF), romiplostim, eltrombopag) must not be used as they may be associated with spleen size increases. Growth factors must not have been used for at least one month prior to receiving the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) | Average of 6 months
  Maximum Tolerated Dose (MTD) of Ruxolitinib with fixed dose of Nilotinib. Dose escalation will follow a 3+3 study design. The CTCAE v4.03 criteria will be used. Grade 4 toxicity will be accounted as dose limiting toxicity (DLT).
Phase II: Major cytogenetic response | Average of 6 months
  Major cytogenetic response defined by 35% or less of Philadelphia chromosomes by metaphase cytogenetics in marrow from CML and ALL patients

SECONDARY OUTCOMES:
Phase I: complete hematologic response | Average of 3 months
  Complete hematologic response defined by CBC differential without any evidence of leukemia. It will be evaluated in CML patients in AP or BP, and patients with Ph+ ALL.
Phase I: major cytogenetic response | Average of 6 months
  Major cytogenetic response defined by 35% or less of Philadelphia chromosomes by metaphase cytogenetics in marrow taken at 6 months.
Phase I: Safety and tolerability | Average of 6 months
  It will be defined by NCI Common Terminology Criteria for Adverse Events (CTCAE)version 4.03 for adverse event reporting.
Phase II: complete hematologic response | Average of 3 months
  Complete hematologic response defined by CBC differential without any evidence of leukemia. It will be evaluated in the CML patients in AP or BP and in patients with Ph+ ALL.

OTHER OUTCOMES:
Phase II (exploratory): pharmacokinetic profile of combination of Nilotinib with Ruxolitinib | During first 24 hours of first dose
  Cmax will be measured for the maximum plasma concentration of nilotinib after oral administration.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Kim, MD/PhD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital / University Health Network, Toronto, Ontario, Canada